CLINICAL TRIAL: NCT00288756
Title: The V-Tachogram:Decreasing Ventricular Arrythmias When Injecting Contrast in the Left Ventricle
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Trillium Health Centre (Other)
Other Study IDs: 01
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2006-09-13 (Estimated); Status verified 2006-09

CONDITIONS: Ventricular Arrythmias
Keywords: arrythmias

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: lv injection of contrast

SUMMARY:
The purpose of this study is to determine if increasing the linear rise rate of injection of x-ray contrast in the heart during left ventriculograms(part of a cardiac Catheterization procedure) will decrease the incidence of arrythmias and improve image quality?

DETAILED DESCRIPTION:
The LV angiogram is performed frequently as part of the cardiac catheterization procedure. It is done by injecting a bolus of x-ray contrast into the ventricle through a pigtail catheter over a short period of time and observing the heart as it is pumped out. This provides information on regional wall motion abnormalities, ejection fraction, and mitral regurgitation. A common occurrence when performing a LV angio is frequent PVC's or V-tach during the injection, it has been suggested that ectopic's occurs about 54% of the time and that interpretability was limited 30% of the time(3) This is rarely serious and subsides at the end of the injection but the irregularity of the contractions does affect the diagnostic quality of the exam.

In an attempt to decrease the incidence of ventricular ectopic's during the LV angiogram Contrast injections with a greater linear rise increasing the injection duration to at least ½ the flow rate, greater than previous settings should decrease the tension and the contrast jets coming out of the catheter, decreasing the fling of the catheter at the initiation of the injection. Whether this affects the quality of the angiogram with a pig tail vs. a straight catheter will also need to be considered?

ELIGIBILITY:
Inclusion Criteria:

* Only ventriculograms that the operator deems necessary for the booked procedure will be considered. Only operators agreeing to the for mentioned settings will participate in the study. Patients will be randomized consecutively and should conclude in 3 to 4 weeks.

Exclusion Criteria:

* Patients with aortic valve disease, a-fib, and frequent benign ectopic beats and patients unable to follow instructions to stop breathing will be excluded.

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156
Dates: Start 2006-07; Study Completion 2006-08

CONTACTS AND LOCATIONS:
Overall Officials: Peter Vandermyden, RN, Principal Investigator — staff RN Trillium Health Centre
Locations (1):
- Trillium Health Centre, Mississauga, Ontario, Canada